CLINICAL TRIAL: NCT03196037
Title: Feasibility of an 8-week Tai Chi Chuan Intervention for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC 1640; 2KR871712 (Other Grant/Funding Number: North Carolina Translational and Clinical Sciences Institute)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Cancer, Breast; Cognitive Impairment
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: A single-arm pre-/post-test non-randomized study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi (Experimental): The Tai Chi intervention will be lead by an expert Tai Chi instructor with 15 years of teaching experience, and will take place at a local Yoga studio. The 8-week intervention entails two 75-minute sessions per week for a total of 16 sessions. Each session will begin with a 15- minute warm-up followed by 25 minutes of performing basic stances, footwork, upper-body/arm/hand movement, proper body alignment, mental/visual focus, and balance; 30 minutes of instruction in a choreographed form (first section of the Yang style long-form); and ending with a 5-minute cool-down.
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Tai Chi — An 8-week Tai Chi intervention consisting of 75-minute group sessions held twice a week, over 8 weeks (i.e., total of 16 sessions).

SUMMARY:
Purpose:To gather preliminary data and to determine the feasibility and acceptability of an 8-week Tai Chi intervention for adults cancer survivors (survivors) who report experiencing cognitive impairment, and to perform exploratory analyses to assess improvements in cognitive performance, health-related quality of life, brain activity, and blood-based biomarkers.

Participants: Adult survivors (> 18 years old) who report experiencing cognitive impairment and are within 60 months of completion of chemotherapy for treatment of a breast cancer diagnosis.

Procedures (methods): A single arm pre-/post-test non-randomized study design in adult cancer survivors (Enrollment goal N=15; current age ≥ 18 years, treatment completed within 60 months). Outcomes will be assessed at baseline and after the 8-week Tai Chi intervention, and consist of feasibility, acceptability, expectancy/credibility, health-related quality of life, cognitive performance, serum biomarkers, and brain activity.

DETAILED DESCRIPTION:
The objective of this study is to gather preliminary data and to determine the feasibility and acceptability of an 8-week Tai Chi intervention for adults within 60 months of having completed chemotherapy for treatment of a cancer diagnosis who report experiencing cognitive impairment (cancer-related cognitive impairment; CRCI). Tai Chi is a form of physical activity that includes an inherent level of cognitive engagement into its performance. Rodent studies provide evidence that including a cognitive component to physical activity (PA) changes its effect on the brain, with aerobic PA inducing angiogenesis and cognitively engaging PA inducing synaptogenesis. Human research with older adults indicates that interventions that combine PA and cognitive engagement produce greater cognitive benefits than PA alone. Experimental and meta-analytic evidence have shown that participation in PA improves cognitive performance in nonclinical and clinical populations, including breast cancer survivors. Importantly, physical activity benefits the same cognitive domains that are negatively affected by CRCI (i.e., attention/processing, memory, executive function). Recently, meta-analytic evidence showed that PA might benefit CRCI. However, in most studies cognitive outcomes are limited to measures of subjective cognitive function rather than objective measures of performance such as neuropsychological assessments or brain activity (e.g., EEG). Research into the effects of Tai Chi on CRCI is sparse, yet promising.

Additionally, research has shown positive effects from Tai Chi on health-related quality of life and cytokines in cancer survivors. To achieve our objective of examining feasibility and acceptability of an 8-week Tai Chi intervention, we will use a single arm pre-/post-test non-randomized study design in adult breast cancer survivors (Enrollment goal N=15; current age ≥ 18 years, treatment completed within 60 months). Outcomes will be assessed at baseline and after the 8-week Tai Chi intervention, and consist of feasibility, acceptability, expectancy/credibility, health-related quality of life, cognitive performance, serum biomarkers, and brain activity. This feasibility study will help identify barriers to recruitment and retention, determine the acceptability of a 8- week Tai Chi intervention for cancer survivors, and provide data for use in designing subsequent studies. Specifically, the findings will inform the design of a randomized controlled trial (RCT) that is sufficiently powered to examine efficacy. The ultimate goal of this research is to create and test a method of investigation into the use of Tai Chi to prevent or mitigate CRCI as well as a method of improving health-related quality of life in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Was diagnosed with breast cancer (all stages accepted).
* Currently > 18 years of age
* Age at cancer diagnosis > 18 years.
* Able to engage in moderate intensity exercise as determined by their treating physician. If participant no longer has a treating physician, safety will be determined by following the American College of Sports Medicine (PAR-Q & YOU) physical activity questionnaire. An answer of "yes" to > one of the seven questions will require the participant to receive written permission from their physician prior to beginning the Tai Chi intervention.
* Not previously engaged in regular exercise training (>1-2d/wk for >30 min/d) in past 6 months.
* Completed chemotherapy treatment for a breast cancer diagnosis.
* Cancer chemotherapy treatment completed within last 60 months. Defined as not currently scheduled for or undergoing active treatment (chemotherapy, radiation, surgery). Treatments to prevent or delay recurrence (e.g., breast cancer hormonal therapies) or for maintenance of remission are allowed.
* Report experiencing cognitive impairment following treatment for cancer.
* No psychiatric disorder with psychotic features.
* Able to receive emails from study staff (i.e. for receiving study reminders).
* Able to speak and read English.
* Able to provide informed consent.

Exclusion Criteria:

* Unwilling or unable to complete study procedures.
* Currently participating in another study which would preclude participation in this study.
* Has a known additional malignancy that is metastatic, progressing, or requires active treatment.
* Has a neurocognitive disorder of other etiologies, such as Alzheimer's Parkinson's, etc., that might confound the analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Feasibility - Attendance | post 8-week intervention
  Feasibility will be achieved if we observe at least 80% attendance (i.e., at least 13 out of 16 sessions attended).
Feasibility Pre-Test Completion | Baseline
  Feasibility will be achieved if we observe at least 80% completion. Completion rates will be the proportion of completed measures (number completed measures/total administered measures at pre-test).
Feasibility Post-Test Completion | post 8-week intervention
  Feasibility will be achieved if we observe at least 80% completion. Completion rates will be the proportion of completed measures (number completed measures/total administered measures at post-test).

SECONDARY OUTCOMES:
Recruitment - Frequency Approached for Screening | Baseline
  We will describe the frequency approached for screening.
Recruitment - Proportion of Completed Screening | Baseline
  We will describe the proportion of completed screening (out of approached for screening)
Recruitment - Screened Eligible | Baseline
  We will describe those screened and found to be eligible (out of total screened).
Retention Rate | post 8-week intervention
  We will describe study retention (number who remain enrolled over 8 weeks/total number originally enrolled).
Recruitment - Enrollment Refusal | Baseline
  We will collect reasons for enrollment refusal (as part of the screening survey)
Retention - Withdrawals | post 8-week intervention
  We will collect reasons for study withdrawals.
Feasibility of the Different Recruitment Strategies - Screened | Baseline
  For each recruitment strategy, we will describe the frequency screened,
Feasibility of the Different Recruitment Strategies - Screened Eligible | Baseline
  For each recruitment strategy, we will describe those screened and found to be eligible (out of total screened).
Feasibility of the Different Recruitment Strategies - Enrolled | Baseline
  For each recruitment strategy, we will describe those enrolled (out of total screened eligible).
Expectancy/Credibility | Baseline
  The Expectancy/Credibility Questionnaire will be used to assess baseline expectancy and credibility effects of taking part in the Tai Chi intervention. Responses to six questions will be indicated with a 1 to 9 Likert-type scale, with higher numbers representing greater expectancy/credibility.
Acceptability | post 8-week intervention
  The Intervention Satisfaction Scale questions: 1) "Overall, I really enjoyed the Tai Chi intervention" and 2) "I would recommend the Tai Chi intervention to other cancer survivors" will assess acceptability. Acceptability will be achieved if the mean score is 3 or greater (response range: 0=Strongly disagree to 4=Strongly agree).
Intervention Satisfaction Questionnaire | post 8-week intervention
  Three close-ended questions will use a Likert scale (0= strongly disagree to 4=strongly agree) to assess whether the class length, frequency, and duration was satisfactory. Four open-ended questions will collect information on what participants liked or disliked about the Tai Chi intervention, and recommendations for changes to better address cancer survivors' needs and basic study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T Piepmeier, PhD, Study Director — University of Rhode Island
Locations (1):
- UNC Chapel Hill Program on Integrative Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan.